CLINICAL TRIAL: NCT00315679
Title: A Trial of Pentoxifylline for the Treatment of Recurrent Aphthous Stomatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHT01
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Recurrent Aphthous Stomatitis
Keywords: recurrent aphthous stomatitis; recurrent mouth ulcers; pentoxifylline; clinical trial; double blind; placebo controlled; randomized
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline (also known as oxpentifylline)

SUMMARY:
This is a randomized, double blind, placebo controlled trial of the use of pentoxifylline (oxpentifylline) for the treatment of recurrent mouth ulcers.

DETAILED DESCRIPTION:
There are few effective treatments for recurrent aphthous stomatitis (cancer sores, recurrent mouth ulcers). Most existing treatments are palliative topical treatments. Some systemic drugs e.g. steroids and thalidomide can suppress the recurrence of mouth ulcers but have serious long term side effects. Pentoxifylline (also known as oxpentifylline) has been used systemically for many years to treat peripheral vascular disease and has a good side effect profile. It shares several actions with thalidomide but does not share its serious side effects. Furthermore, some small scale, open label clinical studies have indicated it may be very effective in treating recurrent aphthous stomatitis (RAS). This study enrolled patients with RAS for which no underlying cause could be identified. Patients kept a diary of the pattern of their mouth ulcers for 60 days to confirm the pattern of ulceration and provide baseline data. Those still qualified for the study were then randomized to treatment with pentoxifylline 400mg three times daily or an identical placebo tablet three times daily for a further 60 days during which they continued to keep a daily ulcer diary. At the end of this period, treatment was stopped and they kept the daily ulcer diary for a further 60 days to identify if any benefit from the treatment was continued after ceasing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of minor recurrent aphthous stomatitis
* 2 or more mouth ulcers per month for more than 6
* No current treatment for oral ulceration or willing to stop treatment
* Age 16 to 65 years

Exclusion Criteria:

* Taking ketorolac, theophylline or anti-hypertensive medication except diuretics (contra-indicated in patients treated with pentoxifylline)
* Systemic diseases that contra-indicate the use of pentoxifylline i.e. pregnancy, hypotension, ischaemic heart disease, acute myocardial infarction, cerebral or occular hemorrhage, renal or hepatic failure, porphyria or allergy to pentoxifylline.
* Patients with an underlying deficiency state or systemic disease that could cause recurrent mouth ulcers e.g. iron, vitamin B12 or foliate deficience, coeliac disease, Crohn's disease, ulcerative colitis, Behcet's disease or Aids.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1996-06; Primary Completion 1998-11 (Actual); Study Completion 1998-11 (Actual)

PRIMARY OUTCOMES:
Reduction in the median pain score
Reduction in the median ulcer size
Reduction in the median ulcer number
Reduction in the total number of episodes of ulceration (RAS)

SECONDARY OUTCOMES:
Change in global ulcer severity score
Increase in the proportion of ulcer free days
Difference in the proportion of ulcer free days (comparing trial v baseline)
Side effect incidence
Side effect type

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Thornhill, MBBS, BDS, Principal Investigator — University of Sheffield School of Clinical Dentistry
Locations (1):
- University Dental Hospital of Manchester, Manchester, United Kingdom

REFERENCES:
- [Derived] Thornhill MH, Baccaglini L, Theaker E, Pemberton MN. A randomized, double-blind, placebo-controlled trial of pentoxifylline for the treatment of recurrent aphthous stomatitis. Arch Dermatol. 2007 Apr;143(4):463-70. doi: 10.1001/archderm.143.4.463. PMID 17438178